CLINICAL TRIAL: NCT07009691
Title: Heart Rate Variability as an Autonomic Marker of Improvement in ME/CFS in a Hydrogen Water Treatment Study
Brief Title: Hydrogen Water Intervention With Heart Rate Variability as an Outcome Biomarker in ME/CFS
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Stony Brook University (Other)
Responsible Party: Principal Investigator, Fred Friedberg, Principal Investigator, Stony Brook University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB2025-00017
Record Dates: First submitted 2025-06-03; First posted 2025-06-08 (Actual); Last update posted 2025-06-08 (Actual); Status verified 2025-06

CONDITIONS: Chronic Fatigue Syndrome
Keywords: Chronic fatigue syndrome; heart rate variability; treatment; hydrogen water.
MeSH Terms: conditions — Fatigue Syndrome, Chronic

STUDY DESIGN:
Intervention Model Description: This is a study of hydrogen water as an intervention for ME/CFS that includes heart rate variability as a potential outcome marker of improvement/non-improvement.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Hydrogen water standard dosage (Experimental): The intervention is hydrogen water which is prepared from an OTC supplement. Hydrogen water is a strong anti-oxidant.
  Interventions: Dietary Supplement: Hydrogen water which is prepared from an OTC supplement.

INTERVENTIONS:
Dietary Supplement: Hydrogen water which is prepared from an OTC supplement. — The intervention is hydrogen water which is prepared from an OTC supplement. It involves measurement of heart rate variability.

SUMMARY:
The goal of this clinical trial is to learn if the OTC supplement, hydrogen water, works to treat the fatigue-related symptoms and functional limitations in adults with myalgic encephalomyelitis/chronic fatigue syndrome (ME/CFS). It will also examine if heart rate variability (HRV) can be used to predict who will benefit from the hydrogen water treatment. The main questions it aims to answer are:

Does the OTC supplement, hydrogen water, work to reduce the fatigue-related symptoms and improve functioning in participants who have ME/CFS?

Can HRV be used to predict who will benefit from treatment with hydrogen water?

DETAILED DESCRIPTION:
The purpose of this pilot study is to identify a biomarker for improvement in chronic fatigue syndrome. Treatment of ME/CFS starting on 10-day graduated dosing schedule followed by a standard daily dose of hydrogen water (a magnesium-based OTC supplement) over 16 weeks is expected to yield two subgroups, improvers and non-improvers. These subgroups will be delineated by heart rate variability (HRV), a biological measure of health and well-being. Higher HRV will predict improvement and lower HRV will predict non-improvement (no change or worsening). This would be the first biomarker of improvement found in ME/CFS. If treatment is successful, subjects will experience a reduction in fatigue and an increase in physical function. Thus, the study may advance potentially an effective intervention for individuals with ME/CFS and further the understanding of the biology of favorable treatment outcomes, i.e., improved HRV status.

ELIGIBILITY:
Inclusion Criteria: Meets Institute of Medicine criteria for myalgic encephalomyelitis/chronic fatigue syndrome -

Exclusion Criteria: Medical illness that explains presenting fatigue; Any psychosis.

-

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2025-06-09 (Estimated); Primary Completion 2026-05-31 (Estimated); Study Completion 2026-05-31 (Estimated)

PRIMARY OUTCOMES:
Fatigue Severity Scale | 12 months
  This is a validated self-report measure of the effect of fatigue on functioning.

CONTACTS AND LOCATIONS:
Overall Officials: Fred Friedberg, PhD, Principal Investigator — Stony Brook University
Locations (1):
- Stony Brook University, Stony Brook, New York, United States